CLINICAL TRIAL: NCT03101176
Title: Multiparametric Ultrasound (mpUS) as Imaging Modality for the Detection and Localization of Prostate Cancer
Brief Title: Multiparametric Ultrasound Imaging in Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prof. dr. ir. H. Wijkstra, prof. dr. Ir. Hessel Wijkstra, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL58710.018.07
Record Dates: First submitted 2017-03-23; First posted 2017-04-05 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer; Prostatic Neoplasms
Keywords: multiparametric ultrasound; prostate cancer; contrast ultrasound; CEUS; radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — contrast agent BR1; Sulfur Hexafluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Single Arm (Experimental): All consenting patients will undergo mpUS imaging prior to surgery with the ultrasound contrast agent Sonovue for the CEUS specific mode.
  Interventions: Drug: SonoVue

INTERVENTIONS:
Drug: SonoVue — The ultrasound contrast agent used for the CEUS specific ultrasound mode
  Other Names: sulphur hexafluoride

SUMMARY:
Rationale: The current limitations in prostate cancer diagnostics, due to lack of accuracy of the available techniques, lead to over- and undertreatment for a significant fraction of patients with prostate cancer. Multiparametric ultrasound (mpUS), a new imaging modality combining different ultrasound parameters, heralds the potential for an accurate imaging-based diagnostic approach accessible to the community at large but formal validation of mpUS against final pathology results are still lacking.

Objective: To validate mpUS as imaging modality for detection and localization of prostate cancer by direct correlation with histopathology of radical prostatectomy specimens

DETAILED DESCRIPTION:
Systematic transrectal ultrasound (TRUS)-guided biopsies in men with a clinical suspicion of prostate cancer, based on digital rectal examination (DRE) and/or prostate-specific antigen (PSA) has been the diagnostic strategy for years. However, this method has known limited sensitivity and risks, as many men without cancer undergo unnecessary biopsies, clinically insignificant cancers are often detected while significant cancers are missed or under-graded and the biopsy procedure itself carries discomfort and morbidity. Prostate imaging capable of identifying clinically significant disease for targeted biopsy with high accuracy and efficiency is thus of importance. mpMRI (multiparametric magnetic resonance imaging) and mpMRI-targeted biopsies are being increasingly used, and they have improved the ability to detect clinically significant cancers, while reducing the diagnosis of insignificant cancers compared to TRUS-guided biopsies. Nevertheless, mpMRI has been limited by inter-reader variability, high level of expertise requirements and heterogeneity in definitions while mpMRI-targeted biopsies alone still misses clinical significant cancers revealed by TRUS-guided biopsies.

There is an ongoing search for new cost-effective, manageable imaging technologies for adequate prostate cancer diagnosis. Various ultrasound modalities are in development striving to increase cancer detection among which contrast-enhanced ultrasound (CEUS) and elastography. Preliminary results of a multiparametric ultrasound (mpUS) approach, combining these different ultrasound modalities, seem promising. The number and quality of studies available, however, is relatively low, emphasizing the need for further work to define the role of mpUS.

This is an investigator-initiated, prospective in-vivo validation study in humans to validate mpUS as imaging modality for detection and localization of prostate cancer by direct correlation with histopathology. Biopsy-proven prostate cancer patients scheduled for radical prostatectomy will be approached and consented to enter this study. Information about the study will be provided both verbally and in written form.

Participants will undergo a mpUS imaging prior to their surgery. For the contrast enhanced mode of the mpUS an additional infusion of an ultrasound contrast agent through an intravenous cannula will be used during transrectal ultrasound scanning for the purpose of the study.

The mpUS imaging data will be evaluated qualitatively and semi-quantitatively using parametric maps by prostate ultrasound experts blinded for radical prostatectomy histopathology. Histopathology will be evaluated qualitatively by an uro-pathologist blinded for mpUS imaging results. Hence, imaging data will be correlated with histopathology in a blinded fashion using a 3D registration system and 3D reconstruction model. Predictive accuracy of mpUS imaging for detection and localization of prostate cancer on histopathology will be analyzed.

At a later stage, a mpUS classifier, most optimally combining the most relevant ultrasound parameters of each modality in one single resulting mpUS parameter will be developed. Furthermore, the additional clinical value of mpUS imaging in prostate cancer diagnostics will be determined by comparing mpUS results with that of available mpMRI data. mpMRI imaging data will be evaluated by an uro-radiologist using the PI-RADS (Prostate Imaging Reporting and Data System) criteria blinded for radical prostatectomy results.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* biopsy proven prostate carcinoma
* planned treatment by (robot laparoscopic) radical prostatectomy
* signed informed consent

Exclusion Criteria:

* Chemotherapy, radiotherapy or focal therapy of the prostate for prostate cancer
* Hormonal therapy for prostate cancer within last six months
* History of any clinically evidence of cardiac right-to-left shunts
* Receives treatment that includes dobutamine
* Severe pulmonary hypertension (pulmonary artery pressure >90 mmHg) or uncontrolled systemic hypertension or respiratory distress syndrome
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study
* Is incapable of understanding the language in which the information for the patient is given

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-09-07 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Validation of mpUS | 5 years
  Predictive accuracy in terms of sensitivity and specificity of mpUS imaging in the detection and localization of prostate cancer by qualitatively and semi-quantitatively correlation of mpUS imaging to corresponding radical prostatectomy histopathology

SECONDARY OUTCOMES:
Differences in mpUS parameters between benign and malignant (low-grade and high-grade) prostate tissue | 5 years
  Parameters of mpUS (echogenicity, contrast-agent perfusion, contrast-agent dispersion, contrast-agent velocity, tissuedensity) will be assessed
mpUS and mpMRI comparison | 5 years
  Comparison of predictive accuracy in terms of sensitivity and specificity of mpMRI imaging and mpUS imaging

CONTACTS AND LOCATIONS:
Overall Officials: H. Wijkstra, Prof dr ir, Principal Investigator — AMC University Hospital
Locations (1):
- AMC University Hospital, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjurlin MA, Carter HB, Schellhammer P, Cookson MS, Gomella LG, Troyer D, Wheeler TM, Schlossberg S, Penson DF, Taneja SS. Optimization of initial prostate biopsy in clinical practice: sampling, labeling and specimen processing. J Urol. 2013 Jun;189(6):2039-46. doi: 10.1016/j.juro.2013.02.072. Epub 2013 Feb 26. PMID 23485507
- [Background] Ukimura O, Coleman JA, de la Taille A, Emberton M, Epstein JI, Freedland SJ, Giannarini G, Kibel AS, Montironi R, Ploussard G, Roobol MJ, Scattoni V, Jones JS. Contemporary role of systematic prostate biopsies: indications, techniques, and implications for patient care. Eur Urol. 2013 Feb;63(2):214-30. doi: 10.1016/j.eururo.2012.09.033. Epub 2012 Sep 25. PMID 23021971
- [Background] Borghesi M, Ahmed H, Nam R, Schaeffer E, Schiavina R, Taneja S, Weidner W, Loeb S. Complications After Systematic, Random, and Image-guided Prostate Biopsy. Eur Urol. 2017 Mar;71(3):353-365. doi: 10.1016/j.eururo.2016.08.004. Epub 2016 Aug 17. PMID 27543165
- [Background] Schoots IG, Roobol MJ, Nieboer D, Bangma CH, Steyerberg EW, Hunink MG. Magnetic resonance imaging-targeted biopsy may enhance the diagnostic accuracy of significant prostate cancer detection compared to standard transrectal ultrasound-guided biopsy: a systematic review and meta-analysis. Eur Urol. 2015 Sep;68(3):438-50. doi: 10.1016/j.eururo.2014.11.037. Epub 2014 Dec 3. PMID 25480312
- [Background] Muller BG, Shih JH, Sankineni S, Marko J, Rais-Bahrami S, George AK, de la Rosette JJ, Merino MJ, Wood BJ, Pinto P, Choyke PL, Turkbey B. Prostate Cancer: Interobserver Agreement and Accuracy with the Revised Prostate Imaging Reporting and Data System at Multiparametric MR Imaging. Radiology. 2015 Dec;277(3):741-50. doi: 10.1148/radiol.2015142818. Epub 2015 Jun 18. PMID 26098458
- [Background] Branger N, Maubon T, Traumann M, Thomassin-Piana J, Brandone N, Taix S, Touzlian J, Brunelle S, Pignot G, Salem N, Gravis G, Walz J. Is negative multiparametric magnetic resonance imaging really able to exclude significant prostate cancer? The real-life experience. BJU Int. 2017 Mar;119(3):449-455. doi: 10.1111/bju.13657. Epub 2016 Oct 4. PMID 27618134
- [Background] Mottet N, Bellmunt J, Bolla M, Briers E, Cumberbatch MG, De Santis M, Fossati N, Gross T, Henry AM, Joniau S, Lam TB, Mason MD, Matveev VB, Moldovan PC, van den Bergh RCN, Van den Broeck T, van der Poel HG, van der Kwast TH, Rouviere O, Schoots IG, Wiegel T, Cornford P. EAU-ESTRO-SIOG Guidelines on Prostate Cancer. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2017 Apr;71(4):618-629. doi: 10.1016/j.eururo.2016.08.003. Epub 2016 Aug 25. PMID 27568654
- [Background] Grey A, Ahmed HU. Multiparametric ultrasound in the diagnosis of prostate cancer. Curr Opin Urol. 2016 Jan;26(1):114-9. doi: 10.1097/MOU.0000000000000245. PMID 26555694
- [Background] Postema A, Mischi M, de la Rosette J, Wijkstra H. Multiparametric ultrasound in the detection of prostate cancer: a systematic review. World J Urol. 2015 Nov;33(11):1651-9. doi: 10.1007/s00345-015-1523-6. Epub 2015 Mar 12. PMID 25761736